CLINICAL TRIAL: NCT05023213
Title: Evaluating "Warna Warni Waktu"; A Social Media-Based Intervention to Improve Body Image and Wellbeing Among Young Indonesian Women
Brief Title: Evaluating an Social Media Intervention to Reduce Body Dissatisfaction Among Young Indonesian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry); University of Hawaii (Other); Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DSEP_GE
Record Dates: First submitted 2021-08-12; First posted 2021-08-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Body Image
Keywords: body dissatisfaction; body satisfaction; positive body image

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The datasets given to the statistician will be blinded to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warna-Warni Waktu intervention (Experimental): Participants in this condition will be asked to view six, approximately five minute videos (each with a number of associated short, interactive reinforcer activities), at a pace of one video per day, for 6 days.
  Interventions: Behavioral: Warna-Warni Waktu
- Waitlist control condition (No Intervention): These participants will no be contacted during the intervention timeframe.

INTERVENTIONS:
Behavioral: Warna-Warni Waktu — Six videos and eighteen reinforcer activities
  Arms: Warna-Warni Waktu intervention

SUMMARY:
The researchers will conduct a randomised controlled trial to evaluate a social media-based intervention aimed at reducing body dissatisfaction among young Indonesian women between 15 and 19 years old. The intervention (titled Warna-Warni Waktu) consists of six sequential videos that tell a fictional story of a typical Indonesian young woman. The videos address known risk factors for body dissatisfaction and include evidence-based techniques to mitigate body dissatisfaction. In addition, the intervention encompasses 18 short online activities intended to encourage participants to think critically about the messages learnt in the videos and practice applying the lessons in real life.

The primary aim is to evaluate the short-term (immediate and four-week post) impact of the intervention on young Indonesian women. The primary outcome is trait body dissatisfaction. Secondary outcomes include internalisation of societal appearance ideals, mood, appearance-related life engagement, and skin shade satisfaction.

The second aim is to evaluate the effectiveness of the videos individually on eliciting state-based improvements (i.e., improvements in the moment) in body dissatisfaction and mood. This will be a within-group design, whereby only participants in the intervention condition will complete single-item measures of body dissatisfaction and mood immediately before and after watching each episode. Further exploratory analyses are also planned.

Approximately 1800 young Indonesian women will be recruited for this research project.

The study's hypotheses are as follows:

1. Participants randomised to the intervention condition will experience reduced body dissatisfaction, skin shade dissatisfaction, and internalisation of appearance ideals, as well as improvements in appearance-related life engagement and mood, at post-intervention, and one-month follow-up, relative to the waitlist control condition.
2. Each video in the Warna-Warni Waktu series will elicit immediate state-based improvements in body satisfaction and mood.
3. Greater engagement and adherence in the Warna-Warni Waktu intervention will result in greater reducing in body dissatisfaction, skin shade dissatisfaction, and internalisation of appearance ideals, as well as improvements in appearance-related life engagement, and mood. This analysis will be exploratory in nature, depending on participants' engagement and adherence in the intervention during the trial.

DETAILED DESCRIPTION:
Background

There is a need for culturally-relevant, accessible, and scalable prevention efforts to reduce body dissatisfaction and improve positive body image among Indonesian girls. Currently, no body image interventions for this population exist.

Recruitment

Participants will be recruited using a local research agency's database of previous research participants.

Previous participants over the age of 40 will be contacted via telephone and screened regarding having a daughter within the eligible age range. If the respondent has more than one daughter in the age range, only one will be eligible. If the respondent does not have a daughter between 15 and 19 years of age, the recruiter will enquire if the respondent knows another family with a daughter of this age. If so, the recruiter will request the telephone number of that family in order to make contact. Only one phone number will be requested per call.

Should an eligible daughter be 15-17 years old, the recruiter will read the parental information sheet to the parent. Parents will then be requested to provide verbal consent for the daughter's participation, as well as verification of the parents' identity and daughter's age. Parents will then answer questions relating to the family's socio-economic status before the recruiter requests to speak to the daughter. If the daughter is not present, the recruiter will request a call back. The daughter will then be screened for eligibility and informed verbal assent obtained. Following a successful call, the parental information sheet will be sent to the parent via WhatsApp, and written informed parental consent obtained.

Should an eligible daughter be aged 18 or 19 years old, a similar pattern of communication will occur. Parents will verify the age of the parents and the daughter, and respond to questions regarding the family's socio-economic status. Rather than parents providing informed verbal and written consent, this will be completed by the daughters, in the same manner with which it will be completed by parents of those aged 15-17 years. Verification of identities and ages will be achieved through video calls via the presentation of a National ID card and family registration card.

Intervention

The intervention, Warna-Warni Waktu (translation to English: Colourful Time Travel), was developed over a 20-month period, from October 2019 - May 2021. In addition to the close collaboration amongst body image academics, creative agencies, social media specialists, not-for-profit organisations, as well as industry funders, development involved three rounds of feedback from the intervention's target audience.

The narrative story told in the six-video series is based on the concept of time travel so as to convey the additive impact of body image concerns to young people. A combination of both animated characters and real people was used.

Four risk factors for the development of body image concerns were identified by the researchers as relevant: 1) social media and influencers 2) appearance-based comparisons 3) appearance-based teasing, and 4) body talk. Each of these risk factors were targeted in videos two through five, with videos one and six being the introductory and concluding videos. Each video is four to five minutes in length. A number of change techniques (including those based upon psychoeducation and media literacy) were embedded within the videos.

Each video is accompanied by one to five short interactive activities, designed to elicit cognitive dissonance. Research consistently shows body image interventions that are interactive generate the most positive outcomes.

Procedure

All participants will enter the study (i.e., complete the baseline assessment questionnaire) on the same day (Day 1). Participants will receive a data package a day prior to this from the research agency to ensure participants have ample mobile phone data to allow participation in the study. A link to the baseline assessment, hosted on Qualtrics (Qualtrics, Provo, UT), will be sent to participants via WhatsApp, along with a unique participant identification number (PIN). Participants will be requested to enter the PIN on the first page of the baseline survey, in order to match participant responses over time. Participants will have 24 hours to complete the baseline assessment; participants that have not completed the baseline assessment within the first 8 hours will be sent a reminder message. Following the 24-hour window, participants who have completed the baseline assessment will be randomised into one of the two conditions. Participants will be alerted on Day 2 to what happens next, depending on which condition each has been randomised. Participants randomised to the intervention condition will be informed to expect a series of links to be sent over the following six days. Participants in the control condition will be informed that contact will be made again in one weeks' time to complete a second assessment.

On the third day (Day 3), participants in the intervention condition will be sent the unique PIN and a link to the first video in the intervention. Again, participants will be requested to enter the unique PIN on the first page of the link. Before watching video one in the Warna-Warni Waktu series, participants will complete state measures of body satisfaction and affect. State measures of body satisfaction and affect will be asked again, immediately after the video. Next, participants will be presented with the reinforcer activities for video one to complete. This process is repeated on Days 4-8, for videos two-six.

On Day 9 of the study, participants in both conditions will be sent a link to complete the second assessment. As with the baseline assessment, participants will be given 24 hours to complete this assessment, with reminder messages sent to non-completers after the first eight hours. The same process will be executed for the third and final assessment, one month later on Day 37.

Following the third assessment, all participants will be debriefed on the study aims and provided with additional sources of mental health support, as well as a certificate of participation. Those in the waitlist control condition will be provided with a link to the Warna-Warni Waktu video series to watch if desired.

ELIGIBILITY:
Inclusion Criteria:

* identifying as a girl
* aged between 15 and 19 years old
* own their own mobile phone
* access Facebook or Instagram daily.

Exclusion Criteria:

* follow the Girl Effect brand ('Springster') on any social media site
* have ever accessed the Springster website
* if under 18 years of age, do not have the written consent from a parent or guardian.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligibility will be determined based on an individual identifying as female.
Enrollment: 1857 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Change in body esteem | baseline; post-intervention (day after the intervention is complete); follow-up (4 weeks later)
  Body esteem will be assessed using the Body Esteem Scale for adolescents & adults (Mendelson, Mendelson & White, 2001), which will be newly validated among Indonesian adolescents prior to the trial. Once the appropriate items are reverse coded, scores on all items are averaged; with lower scores indicating lower body esteem.

SECONDARY OUTCOMES:
Change in internalisation of societal appearance ideals | baseline; post-intervention (day after the intervention is complete); follow-up (4 weeks later)
  Internalisation of societal appearance ideals will be assessed using The Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3): General Subscale, newly validated among Indonesian adolescents. Scores are averaged, with higher scores indicating higher internalisation.
Change in mood | baseline; post-intervention (day after the intervention is complete); follow-up (4 weeks later)
  Positive and Negative affect will be measured using the Positive and Negative Affect Schedule (Crawford & Henry, 2004), newly validated among Indonesian adolescents. Scores on each subscales are averaged; with higher scores indicating greater negative affect and positive affect respectively.
Change in life engagement | baseline; post-intervention (day after the intervention is complete); follow-up (4 weeks later)
  Opting out of important life activities due to body image concerns will be assessed using the Body Image Life Engagement Questionnaire (BILEQ; Atkinson & Diedrichs, 2021), newly validated among Indonesian adolescents. This measure assesses the extent that worries or feeling bad about the way you look has stopped you, or are likely to stop you, from engaging in life activities (e.g., going to a social event, doing physical activity, giving an opinion, going to school). Scores on all items are averaged; with higher scores indicating greater avoidance of activities due to appearance concerns.
Change in skin shade satisfaction | baseline; post-intervention (day after the intervention is complete); follow-up (4 weeks later)
  Single-item, purpose built measure to assess satisfaction with skin shade.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Garbett, MSc, Principal Investigator — University of the West of England
Locations (1):
- University of the West of England, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garbett KM, Craddock N, Haywood S, Nasution K, White P, Saraswati LA, Medise BE; Girl Effect; Percolate Galactic; Diedrichs PC, Williamson H. A Novel, Scalable Social Media-Based Intervention ("Warna-Warni Waktu") to Reduce Body Dissatisfaction Among Young Indonesian Women: Protocol for a Parallel Randomized Controlled Trial. JMIR Res Protoc. 2022 Jan 28;11(1):e33596. doi: 10.2196/33596. PMID 35089154